CLINICAL TRIAL: NCT01268917
Title: The Effects of Preoperative Aspirin on Graft Patency and Cardiac Events in Off-pump Coronary Artery Bypass
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Fuwai Hospital, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fuwai Hospital 2010-259
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Disease; Off-pump Coronary Artery Bypass; Aspirin
Keywords: coronary artery disease; off-pump coronary artery bypass; aspirin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- preoperative aspirin use (Experimental)
  Interventions: Drug: aspirin
- preoperative aspirin nonuse (No Intervention)
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — aspirin 100mg daily until the surgery day
  Arms: preoperative aspirin use
Drug: aspirin — aspirin is stopped 5-7 days before operation
  Arms: preoperative aspirin nonuse

SUMMARY:
Antiplatelet therapy is critical in the management of coronary artery disease.For patients undergoing off-pump coronary artery bypass graft,controversy remains regarding the safety of preoperative antiplatelet therapy.And there is little study about the effect of continuing aspirin until the surgery day on graft patency.So we would like to perform this study to evaluate the effects of preoperative aspirin on graft patency and cardiac events in off-pump coronary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective, off-pump coronary artery bypass with at least two grafts
* patient able to give informed consent

Exclusion Criteria:

* on-pump CABG
* combined with the valve surgery
* Preoperative use of clopidogrel and warfarin
* allergy to aspirin
* History of severe liver disease
* History of bleeding diathesis,significant GI bleed
* Patient has known renal failure or contraindication for Cardiac CT Angio
* Redo CABG

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
graft patency examined by CT scan | one week after surgery
  we would like to compare the graft patency within the one week after the surgery between the preoperative aspirin use and preoperative nonuse.We just want to know wether preoperative aspirin use could improve the graft patency in off-pump coronary artery bypass.

SECONDARY OUTCOMES:
Bleeding, transfusion, re-exploration | perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China

REFERENCES:
- [Derived] Chen S, Wu H, Yang T, Li B, Hu Y, Sun H. Does Early Graft Patency Benefit from Perioperative Statin Therapy? A Propensity Score-Matched Study of Patients Undergoing Off-Pump Coronary Artery Bypass Surgery. Cardiovasc Ther. 2019 Aug 6;2019:1582183. doi: 10.1155/2019/1582183. eCollection 2019. PMID 31772605